CLINICAL TRIAL: NCT00723268
Title: Evaluation of Therapeutic Effect of 0.5 mg Colchicine and 5 mg Prednisolone on Oral Aphthae
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: University of Tehran (Other)
Responsible Party: Mashhad University of Medical Science, Mashhad Dental Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 286293; 286293
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Oral Aphthae
Keywords: Oral ulcers
MeSH Terms: conditions — Foot-and-Mouth Disease; Oral Ulcer | interventions — Prednisolone; Colchicine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Active Comparator)
  Interventions: Drug: Prednisolone
- Colchicine (Active Comparator)
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Prednisolone — 5MG Prednisolone per day for 3 months
  Arms: Prednisolone
Drug: Colchicine — 0.5 MG Colchicine per day for 3 months
  Arms: Colchicine

SUMMARY:
The purpose of this study is to determine whether low doses of prednisolone, or colchicine are effective in the treatment of oral aphthae.

DETAILED DESCRIPTION:
Treatment of recurrent aphthous stomatitis (RAS) remains, to date, empirical and non-specific. The main goals of therapy are to minimize pain and functional disabilities as well as decrease inflammatory reactions and frequency of recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of clinical diagnosis of aphthae
* Having the experience of oral aphthae at least once in a month
* Two weeks wash out periods after the last treatment

Exclusion Criteria:

* History of any systemic disease
* Using drugs which affect immune system
* Pregnancy and breast feeding
* Aphthous related syndromes

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
frequency of ulcers | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad Dental school, Mashhad, Khorasan Razavi, Iran